CLINICAL TRIAL: NCT06819111
Title: Kinetics of Urinary Alkalinization Therapy in Patients With Nephrolithiasis
Brief Title: Role of Medication in Making Urine Less Acidic as Part of Kidney Stone Prevention
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Brett Johnson, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU-2024-1257
Record Dates: First submitted 2025-01-27; First posted 2025-02-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Kidney Calculi
Keywords: kidney stone prevention; potassium citrate; urine alkalization
MeSH Terms: conditions — Kidney Calculi | interventions — potassium-magnesium citrate; Powders; Tablets

STUDY DESIGN:
Intervention Model Description: The crossover design of our study was intentional to allow patients to serve as their own controls across multiple study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Urine Alkalization (Experimental): In this crossover study, patients will serve as their own controls. Patients will receive slow-release potassium citrate (UroCit-K), potassium magnesium citrate (powder), or potassium magnesium citrate (tablets). The study period will last approximately 6 weeks for each participant. Patients will be instructed to take one form of potassium citrate for one week at a time followed by a washout period for one week. This process will be completed a total of three times as we seek to study the effects of three forms of potassium citrate.
  Interventions: Drug: Potassium Citrate Extended Release Oral Tablet

INTERVENTIONS:
Drug: Potassium Citrate Extended Release Oral Tablet — In this crossover study, patients will serve as their own controls. Patients will receive slow-release potassium citrate (UroCit-K), potassium magnesium citrate (powder), or potassium magnesium citrate (tablets). The study period will last approximately 6 weeks for each participant. Patients will be instructed to take one form of potassium citrate for one week at a time followed by a washout period for one week. This process will be completed a total of three times as we seek to study the effects of three forms of potassium citrate.
  Other Names: potassium magnesium citrate (powder); potassium magnesium citrate (tablets)

SUMMARY:
Diet and medications are the cornerstones of kidney stone prevention. Potassium citrate is a commonly prescribed medication to help prevent kidney stones by making urine less acidic. There are different forms of potassium citrate such as over-the-counter tablet or powder, and slow-release tablets that require a prescription. However, it is unknown if one form is better than the others. Therefore, we want to compare different forms of potassium citrate and find out how well they work and whether patients prefer one form over the others.

The study period will last approximately 6 weeks for each participant. Patients will be instructed to take one form of potassium citrate for one week at a time followed by a washout period for one week. This process will be completed a total of three times as we seek to study the effects of three forms of potassium citrate.

At the end of each trial week patients will be asked to provide urine samples and complete two surveys. Urine will need to be collected for 24 hours, which will then be examined to determine the effects that each form of potassium citrate has on urine. In addition, completed surveys will give us information on how well the medication was tolerated and their satisfaction with the treatment. There is a possibility that patients like one form better than others, and it is also possible that they do not see a difference at all.

Throughout the duration of the study patients will be asked to be a directed diet. This will be based on general recommendations by the National Kidney Foundation for the prevention of kidney stones.

DETAILED DESCRIPTION:
Background and Rationale

Urinary stone disease (USD) has been increasing with a recent prevalence estimate of 11% in the United States. Recurrence is common, with up to 50% of individuals experiencing another stone event within 10 years without treatment. This condition results in pain, diminished quality of life, missed work and school, as well as chronic kidney disease and renal failure, and carries significant economic implications as USD is the most expensive non-malignant urologic condition in the United States.

Diet modification and pharmacotherapy form the cornerstones of kidney stone prevention. Alkalinization of urine is commonly used to prevent kidney stone recurrence. Physiologically, urine alkalinization increases urinary pH and raises urinary citrate levels. Correction of acidic urine pH (<5.5) can counteract uric acid crystallization. Additionally, increased citrate levels are known to be a potent inhibitor of calcium stone formation by binding directly to urinary calcium and inhibiting crystal nucleation. Therefore, alkali therapy addresses risk factors for several types of kidney stones and is recommended for patients with recurrent calcium stones with or without hypocitraturia, uric acid stones, or cystine stones.

Potassium citrate is the most commonly prescribed form of alkali therapy. It is recommended by multiple national society guidelines for patients with recurrent calcium stones in whom modifiable 24-hour urine (24U) risk factors are absent, already addressed, or for those in whom dietary modification alone was ineffective. Unfortunately, the long-term compliance has been reported to be as low as 13%. Part of the problem is that potassium citrate is not well-tolerated due to its gastrointestinal side effect profile. So even if urinary alkalization is more robust with potassium citrate, the clinical effects will not be realized if patients are not compliant with the medication. Further exacerbating noncompliance is the unavailability of desirable powder forms of potassium citrate (crystal packets), or the cost of the slow-release form of potassium citrate (UroCit-K) estimated to be more than $150 per month, which may be prohibitively expensive for some patients. Additionally, the number of pills needed to be taken on a daily basis is another reason that could lead to noncompliance.

Alternative alkali therapies are available and should be considered. Over-the-counter (OTC) alkali therapy including medicinal foods and dietary supplements have been used as alternatives to traditional potassium citrate therapy for urinary alkalinization. Indeed, OTC therapies are growing in popularity, with half of recurrent stone-formers reporting utilization of alternative medicines. Moreover, the large number of available products further supports the high demand for such alternative agents. However, there is limited evidence to support their use and efficacy as the comparative efficacy, cost, and tolerability between these agents compared to the current gold standard potassium citrate therapy is unknown.

Our research group has previously studied commonly available OTC alternative alkali citrate products to determine the actual quantities of citrate and citrate as alkali in these supplements. This included powder products such as Litholyte®, Moonstone®, and NOW® Potassium citrate. Litholyte® powder was felt to provide reasonable balance between alkali citrate, cost, and ease of consumption. To build upon this work, we aim to perform an open-label Phase-1 clinical trial using Litholyte®, a dietary supplement containing potassium/magnesium citrate, and compare its metabolic effects to the gold standard potassium citrate (UroCit-K) therapy. We hypothesize that in recurrent stone formers, Litholyte® products will result in similar urinary alkalinization and urinary citrate levels compared to UroCit-K but will be better tolerated and less costly.

ELIGIBILITY:
Inclusion Criteria:

* adults, 18 years or older
* recurrent stone formers or first-time stone formers at high risk for recurrence
* have a baseline 24-hour urine within six months from study enrollment
* have the ability to adhere to a directed diet

Exclusion Criteria:

* minors (age <18 years)
* mentally incapacitated and/or unable to provide consent
* prisoners
* pregnant or breastfeeding individuals
* concurrent potassium citrate therapy
* concurrent thiazide therapy
* chronic kidney disease (eGFR <60)
* solitary kidney
* unable to take any of the study medications due to a prior adverse reaction or other health-related reason (ex: severe renal impairment, hyperkalemia, or severe acidosis or alkalosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Urinary pH | From enrollment to the end of treatment at 6 weeks.
  Change in urinary pH and urinary citrate

IPD SHARING:
Plan to Share IPD: No
This is a single center study